CLINICAL TRIAL: NCT05807763
Title: Selective Use of Fundoplication in Laparoscopic Paraesophageal Hernia Repair Based on Intra-operative Impedance Planimetry (FLIP)
Brief Title: Fundoplication in Laparoscopic PEH Repair Based on FLIP
Acronym: PEHFLIP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Foundation for Surgical Innovation and Education (Other)
Responsible Party: Principal Investigator, Christy M. Dunst, Program Director Complex GI-Foregut Fellowship, Providence Portland Medical Center, The Oregon Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY2022000698
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-04

CONDITIONS: Paraesophageal Hernia
Keywords: Paraesophageal hernia repair; Laparoscopic paraesophageal hernia repair; PEH repair; Lap PEH repair; FLIP; Functional luminal imaging probe; GERD; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Fundoplication
- Study Group (Experimental): No Fundoplication
  Interventions: Procedure: Laparoscopic paraesophageal hernia repair without fundoplication

INTERVENTIONS:
Procedure: Laparoscopic paraesophageal hernia repair without fundoplication — Patients undergoing laparoscopic paraesophageal hernia repair will be evaluated for risk of esophageal reflux using intra-operative impedance planimetry and endoscopic gastroesophageal valve grade. Patients deemed low risk for esophageal reflux will then be randomized to "partial fundoplication" or "no fundoplication".
  Arms: Study Group

SUMMARY:
Prospective randomized controlled trial to identify a sub-set of patients that do not benefit from the routine addition, and added morbidity, of a fundoplication during laparoscopic paraesophageal hernia repair.

DETAILED DESCRIPTION:
Prospective Randomized Controlled Trial in which patients who meet criteria will be randomized to receive a concurrent fundoplication or no fundoplication at the time of paraesophageal hernia repair. Patients with known objective gastroesophageal reflux disease prior to surgery, those found to have a short esophagus in the operating room or defective gastroesophageal reflux barrier by intra-operative impedance planimetry measurements and/or endoscopic valve grade will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic paraesophageal hernia repair

Exclusion Criteria:

* History of a prior hiatal hernia/paraesophageal hernia repair
* Patients with objective GERD preoperatively
* Intra-operative short esophagus
* Defective gastroesophageal reflux barrier as determined by impedance planimetry (FLIP)
* Defective gastroesophageal reflux barrier as determined by intra-operative endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-02-22 (Estimated); Study Completion 2029-02-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with GERD post-op | 12 months
  Patients will undergo endoscopic evaluation and 48 hour pH testing to determine the incidence of objective GERD with and without fundoplication after PEH repair.

SECONDARY OUTCOMES:
Number of participants with hernia recurrence | 12 months
  Routine upper GI contrast study and endoscopy will evaluate for hernia recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Christy M Dunst, MD, Principal Investigator — The Oregon Clinic
Locations (2):
- United States (2):
  - NorthShore University HealthSystem, Evanston, Illinois
  - Providence Portland Medical Center / The Oregon Clinic, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller-Stich BP, Achtstatter V, Diener MK, Gondan M, Warschkow R, Marra F, Zerz A, Gutt CN, Buchler MW, Linke GR. Repair of Paraesophageal Hiatal Hernias-Is a Fundoplication Needed? A Randomized Controlled Pilot Trial. J Am Coll Surg. 2015 Aug;221(2):602-10. doi: 10.1016/j.jamcollsurg.2015.03.003. Epub 2015 Mar 14. PMID 25868406
- [Background] Su B, Dunst C, Gould J, Jobe B, Severson P, Newhams K, Sachs A, Ujiki M. Experience-based expert consensus on the intra-operative usage of the Endoflip impedance planimetry system. Surg Endosc. 2021 Jun;35(6):2731-2742. doi: 10.1007/s00464-020-07704-3. Epub 2020 Jun 16. PMID 32556758
- [Background] Wu H, Attaar M, Wong HJ, Campbell M, Kuchta K, Denham EW 3rd, Linn J, Ujiki MB. Impedance Planimetry (Endoflip) and Ideal Distensibility Ranges for Optimal Outcomes after Nissen and Toupet Fundoplication. J Am Coll Surg. 2022 Sep 1;235(3):420-429. doi: 10.1097/XCS.0000000000000273. Epub 2022 Aug 10. PMID 35972160
- [Background] Heard, J, DuPree, C, Ibrahim M, Karumuri J, Osman, H, Jeyarajah, R. Endoflip Driven Paraesophageal Hernia Repair without Fundoplication: Heresy or Good Practice? Abstract accepted for presentation at Society for Surgery of the Alimentary Tract (SSAT) Annual Meeting 2023.
- [Background] Rieder E, Swanstrom LL, Perretta S, Lenglinger J, Riegler M, Dunst CM. Intraoperative assessment of esophagogastric junction distensibility during per oral endoscopic myotomy (POEM) for esophageal motility disorders. Surg Endosc. 2013 Feb;27(2):400-5. doi: 10.1007/s00464-012-2484-0. Epub 2012 Sep 6. PMID 22955896
- [Background] Attaar M, Wong HJ, Wu H, Campbell M, Kuchta K, Denham W, Haggerty S, Linn J, Ujiki MB. Changes in impedance planimetry (EndoFLIP) measurements at follow-up after peroral endoscopic myotomy (POEM). Surg Endosc. 2022 Dec;36(12):9410-9415. doi: 10.1007/s00464-022-09286-8. Epub 2022 May 3. PMID 35505258
- [Background] Wu H, Attaar M, Wong HJ, Campbell M, Kuchta K, Denham W, Linn J, Ujiki MB. Impedance planimetry (EndoFLIP) after magnetic sphincter augmentation (LINX(R)) compared to fundoplication. Surg Endosc. 2022 Oct;36(10):7709-7716. doi: 10.1007/s00464-022-09128-7. Epub 2022 Feb 15. PMID 35169878
- [Background] Amundson JR, Wu H, VanDruff V, Campbell M, Kuchta K, Hedberg HM, Ujiki MB. Esophagogastric junction compliance on impedance planimetry (EndoFLIP) following peroral endoscopic myotomy (POEM) predicts improvement in postoperative eckardt score. Surg Endosc. 2023 Feb;37(2):1493-1500. doi: 10.1007/s00464-022-09432-2. Epub 2022 Jul 15. PMID 35838832